CLINICAL TRIAL: NCT00581334
Title: Robotic-assisted Laparoscopic Sacrocolpopexy: A Feasibility Study
Brief Title: Robotic-assisted Laparoscopic Sacrocolpopexy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Felicia Lane, Professor and Vice Chair of Obstetrics & Gynecology, University of California, Irvine
Other Study IDs: 20054606
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Robotic-assisted laparoscopic sacrocolpopexy; Post hysterectomy prolapse; Symptomatic apical prolapse of stage II or >
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Robotic Sacrocolpopexy Group: laparoscopic mesh augmented prolapse repair for post-hysterectomy prolapse repair using the Da Vinci robot
  Interventions: Procedure: Robotic-assisted laparoscopic sacrocolpopexy
- Open Sacrocolpopexy Group: matched cohort that underwent mesh augmented prolapse repair for post-hysterectomy prolapse performed via open laparotomy
  Interventions: Procedure: Open sacrocolpopexy

INTERVENTIONS:
Procedure: Robotic-assisted laparoscopic sacrocolpopexy — 4 abdominal incisions will be made: 1 infraumbilical port and 3 lateral ports. The peritoneum overlaying the sacrum is entered and the anterior longitudinal ligament is exposed. 3 permanent sutures are placed through the ligament at the S2-S3. Then a vaginal obturator is placed transvaginally and the apex of vagina is elevated into the operative field. The peritoneum overlying the anterior and posterior vaginal epithelium is reflected and the bladder is dissected off the underlying vagina to expose 4cm of apical vagina. 2 segments of polypropylene mesh are prepared and one segment is anchored along the anterior vagina with a series of interrupted permanent suture and the second segment is anchored along the posterior vagina. These 2 segments are brought together to the previously placed sutures within the anterior longitudinal ligament of the sacrum. The peritoneum is then closed over the graft complex and the pelvis irrigated. The 4 robotic ports are removed and the abdomen closed.
  Other Names: DaVinci Robotic System
  Groups: Robotic Sacrocolpopexy Group
Procedure: Open sacrocolpopexy — mesh augmented repair for post-hysterectomy prolapse performed via open laparotomy
  Groups: Open Sacrocolpopexy Group

SUMMARY:
Robotic-assisted Abdominal Sacrocolpopexy is both a feasible and safe method for apical prolapse repair of the vagina.

DETAILED DESCRIPTION:
Robotics offers many advantages over traditional laparoscopy: 1) intuitive movement of instruments, 2) "wristed instruments" with increased degrees of freedom, 3) enhanced 12X magnification, 4) 3-D depth perception, 5)tremor filtration, 6) enhanced surgeon comfort and ergonomics, and 7) a steeper learning curve. With robotic assistance, the surgeon can comfortably perform precise, repetitive motions, with greater dexterity and vision. To date, there have been a small number of published cases of laparoscopic sacrocolpopexy and two cases of series utilizing robotic-assistance. There have been no prospective, randomized, controlled trials comparing either of these modalities to conventional abdominal sacrocolpopexy.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women
* Age >18 years
* Eligible for sacrocolpopexy
* Prior hysterectomy
* Stage II or greater post hysterectomy vault prolapse
* Satisfied parity
* Patients electing for an abdominal repair to posthysterectomy vault prolapse

Exclusion Criteria:

* Prisoners
* Cognitively impaired adults
* Not medically stable to undergo laparoscopic or abdominal surgery
* Previous pelvic/vaginal radiation
* Participants electing to proceed with a vaginal repair of vaginal vault prolapse
* Participants electing to proceed with the traditional abdominal sacrocolpopexy
* History of recurrent vaginal infections
* Known urologic and/or gynecologic cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gynecology patients undergoing colpopexy.
Study Population: Female urogynecology patient with symptomatic apical prolapse
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are operative time, blood loss, complication rates, length of hospital stay, and cure. Objective cure can be measured using the pelvic organ prolapse quantification exam (POP-Q). | 2 years
  time, estimated blood loss, UTI, duration-of stay

SECONDARY OUTCOMES:
Secondary outcomes will measure the effects of the surgical repair using a series of questionnaires: SF-36, Pelvic Floor Distress Inventory which includes Pelvic Organ Prolapse Impact, Colo-Rectal-Anal Impact, and Urinary Impact Questionnaire. | 2 Years
  validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States